CLINICAL TRIAL: NCT03550508
Title: A Phase I, Multi-center, Open-label, Dose Escalation Study to Evaluate the Safety, Tolerability and Preliminary Pharmacokinetics/Pharmacodynamics of JMT103 in Patients With Bone Metastases From Tumors
Brief Title: Safety, Tolerability and PK/PD of JMT103 in Patients With Bone Metastases From Tumors
Acronym: JMT103
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry); Covance (Industry); KingMed Diagnostics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT103CN01
Record Dates: First submitted 2018-04-18; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Bone Metastases
Keywords: JMT103 in Patients with Bone Metastases from Tumors

STUDY DESIGN:
Intervention Model Description: The accelerated titration and traditional "3+3" dose-escalation designs are applied in this study.
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-RANKL Monoclonal Antibody (Experimental): Anti-RANKL Monoclonal Antibody is to be injected subcutaneously 0.5 mg/kg, 1.0 mg/kg, 2.0 mg/kg or 3.0 mg/kg.
  Interventions: Biological: Anti-RANKL Monoclonal Antibody

INTERVENTIONS:
Biological: Anti-RANKL Monoclonal Antibody — JMT103 is recombinant fully human anti-RANKL monoclonal antibody. JMT103 is provided as the injection,120 mg/vial. JMT103 was administered subcutaneously in the upper arm, upper thigh, or abdomen.
  Other Names: JMT103

SUMMARY:
JMT103 is a novel, full human IgG4 monoclonal antibody targeting RANKL. In preclinical studies, JMT103 demonstrated strong activity through blocking RANKL receptor, RANK on the surface of osteoclasts, leading to inhibit osteoclast differentiation, activation, and maturation and reduce bone resorption.

This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) ,to evaluate the safety, pharmacokinetics and preliminary efficacy (bone turnover markers) of recombinant fully human Anti-RANKL Monoclonal Antibody (JMT103) in patients with bone metastases from tumors at single doses and multiple doses.

About 36 cases patients are to be recruited.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, multi-center, open-label dose escalation clinical study of recombinant fully human Anti-RANKL Monoclonal Antibody (JMT103) administered subcutaneously to patients with bone metastases from tumors.

The study includes two phases: dose escalation study and expansion study. The dose-escalation stage is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and following repeat doses of JMT103 given every 4 weeks (Q4W) for three times. The expansion study stage is designed to evaluate the safety, tolerability, and pharmacokinetics of repeat doses of JMT103 given every 4 weeks (Q4W) for three times.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed malignant solid tumors;
* imaging examination shows at least one site with bone metastases from tumors;
* ECOG performance status of score 0 or 1;
* Expected survival time ≥ 7.5 months.

Exclusion Criteria:

* Previous or present osteomyelitis or osteonecrosis of the jaw; unhealed dental or oral surgery wounds; acute disease of the tooth or jaw requiring oral surgery; and invasive dental surgery planned to be received during the study;
* It is planned to perform therapeutic radiotherapy or orthopedic surgery for patients during the study;
* Known active brain metastases or leptomeningeal metastases. The subjects with neurological symptoms should receive brain CT/MRI to ensure that there have no metastases;
* Patients with bone metabolic diseases (Paget's disease, Cushing syndrome and hyperprolactinemia), rheumatoid arthritis, and current hyperparathyroidism or parathyroid dysfunction;
* Uncontrolled complications
* Active bacterial or fungal infections requiring systematic treatment within 7 days before the screening;
* Patients with HIV infections or active hepatitis;
* Pregnancy (positive serum β-HCG result) or lactation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 28 days

SECONDARY OUTCOMES:
Anti-Drug Antibody of Anti-RANKL Monoclonal Antibody (JMT103) in Patients With Bone Metastases From Tumors | 225 days in escalation study stage, and 141 days in expansion study stage
Maximum serum Concentration (Cmax) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Peak Time (Tmax) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Area Under the Curve (AUC) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Terminal t1/2 after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Serum clearance (CL) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Apparent volume of distribution (V) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Minimum serum Concentration (Cmin) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Minimum serum Concentration (Cmin) after multiple dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 141 days
Apparent volume of distribution after multiple dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 141 days
Cumulative factor after multiple dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 141 days
Percent changes of serum C-terminal telopeptide of type 1 collagen after single dose of JMT103 | 85 days
Percent changes of bone alkaline phosphatase after single dose of JMT103 | 85 days
Percent changes of procollagen type 1 N-peptide, tartrate-resistant acid phosphatase 5b (TRAP5b) after single dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 85 days
Percent changes of urinary N-terminal telopeptide of type 1 collagen/creatine (U-NTX/Cr) after multiple doses of JMT103 | 141 days
Percent changes of serum C-terminal telopeptide of type 1 collagen after multiple doses of JMT103 | 141 days
Percent changes of bone alkaline phosphatase after multiple doses of JMT103 | 141 days
Percent changes of procollagen type 1 N-peptide, tartrate-resistant acid phosphatase 5b (TRAP5b) after multiple doses of JMT103 | 141 days
Percent changes of urinary N-terminal telopeptide of type 1 collagen/creatine (U-NTX/Cr) after multiple dose injection of Anti-RANKL Monoclonal Antibody (JMT103) | 141 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang X, Xue J, Ge X, Li J, Li H, Xue L, Di L, Tang W, Song G, Li Q, Jiang H, Zhao W, Lin F, Shao B, Yang X, Wu Z, Zhang T, Wang C, Guo Y. Safety, tolerability, and pharmacokinetics/pharmacodynamics of JMT103 in patients with bone metastases from solid tumors. Front Oncol. 2022 Aug 5;12:971594. doi: 10.3389/fonc.2022.971594. eCollection 2022. PMID 35992822